CLINICAL TRIAL: NCT07212907
Title: Effect of a Combination of Spore-forming Probiotics (Bacillus Coagulans MY01 and Bacillus Subtilis MY02) and Ginger Extract on Symptoms and Quality of Life in Patients With Functional Dyspepsia
Brief Title: Probiotic and Ginger Supplement for Symptoms and Quality of Life in Functional Dyspepsia (SUBTILE)
Acronym: SUBTILE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biocodex (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUBTILE - STO 253; 2025-A01409-40 (Other: IDRCB (France))
Record Dates: First submitted 2025-08-29; First posted 2025-10-08 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-09

CONDITIONS: Functional Dyspepsia
Keywords: Functional Dyspepsia; Bacillus coagulans MY01; Bacillus subtilis MY02; Ginger extract; Symbiosys Stomalex; Gut microbiota; Quality of life; Gastrointestinal symptoms; Spore-forming probiotics; Epigastric Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Single-arm, prospective, multicenter interventional study evaluating a dietary supplement containing Bacillus coagulans MY01, Bacillus subtilis MY02, and ginger extract in patients with functional dyspepsia
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Probiotic and Ginger Supplement (Experimental): Patients with functional dyspepsia will receive one capsule per day of a dietary supplement containing Bacillus coagulans MY01, Bacillus subtilis MY02, and ginger extract (50 mg, 20% gingerols) for 8 weeks
  Interventions: Dietary Supplement: Symbiosys® Stomalex (commercial name)

INTERVENTIONS:
Dietary Supplement: Symbiosys® Stomalex (commercial name) — One oral capsule per day for 8 weeks. Each capsule contains Bacillus coagulans MY01, Bacillus subtilis MY02, and ginger root extract (50 mg, titrated to 20% gingerols).

SUMMARY:
Functional dyspepsia (FD) is a frequent functional gastrointestinal disorder characterized by bothersome postprandial fullness, early satiety, epigastric pain, or burning, in the absence of any structural or metabolic cause. It significantly impairs quality of life and has limited therapeutic options, as conventional treatments such as proton pump inhibitors often show modest efficacy and may cause side effects with long-term use.

The gut and duodenal microbiota may play a role in FD. Spore-forming probiotics such as Bacillus coagulans MY01 and Bacillus subtilis MY02 have shown beneficial effects on FD symptoms in a randomized controlled trial. Ginger (Zingiber officinale) has a long history of traditional use as a gastroprotective agent and is supported by clinical and non-clinical data for improving gastric motility and related symptoms.

This study (SUBTILE, STO-253) is a prospective, interventional, multicenter trial conducted in France. It will evaluate the effect of a dietary supplement containing Bacillus coagulans MY01, Bacillus subtilis MY02, and ginger extract (50 mg, 20% gingerols) on FD symptoms and quality of life.

A total of 198 adult patients diagnosed with FD according to Rome IV criteria and with a normal upper endoscopy will be recruited in primary care and gastroenterology practices. Participants will take one capsule of the study product daily for 8 weeks.

The primary outcome is the change in the Patient Assessment of Gastrointestinal Symptom Severity (PAGI-SYM) total score between baseline and Week 8.

Secondary outcomes include changes in quality of life (PAGI-QoL), treatment adherence, use of concomitant medications, evolution of lower gastrointestinal symptoms, patient and physician global impressions of change (PGI-C, CGI-I), and satisfaction (Likert scales). An exploratory objective will assess psychological impact using the Hospital Anxiety and Depression Scale (HADS).

The study includes two site visits (baseline and end of study) and one telephone follow-up at Day 28. Safety and tolerability will be monitored through active reporting of adverse events.

The trial aims to provide new evidence on the role of probiotics combined with ginger extract as a non-pharmacological strategy to improve digestive comfort and quality of life in patients with functional dyspepsia.

DETAILED DESCRIPTION:
Functional dyspepsia (FD) is one of the most common disorders of gut-brain interaction (DGBI), with an estimated prevalence of 7-8% in the general population. It is defined by Rome IV criteria as bothersome postprandial fullness, early satiety, epigastric pain, or burning, persisting for at least 3 months with onset at least 6 months before diagnosis, and without evidence of structural disease. FD is associated with impaired quality of life, psychological distress, and significant health care utilization. Current treatment options, including proton pump inhibitors and prokinetics, have limited efficacy and potential adverse effects when used long term.

Emerging evidence suggests a role of the gastrointestinal microbiota in FD pathophysiology. Alterations in duodenal microbiota, as well as small intestinal bacterial overgrowth (SIBO) promoted by chronic PPI use, have been reported. Probiotics may reduce dyspeptic symptoms, improve gut barrier function, modulate gastric motility, and exert anti-inflammatory effects.

A randomized controlled trial showed that Bacillus coagulans MY01 and Bacillus subtilis MY02 improved FD symptoms compared to placebo, with good safety and tolerability. In parallel, ginger (Zingiber officinale) has a well-documented gastroprotective effect, supported by both preclinical and clinical data, and has been shown to enhance gastric emptying and reduce upper gastrointestinal discomfort.

The present study (SUBTILE, STO-253) is a prospective, multicenter, interventional trial conducted in France, categorized as RIPH2 (research involving human participants at minimal risks and constraints) under French regulations. The study will evaluate the effect of a dietary supplement combining Bacillus coagulans MY01, Bacillus subtilis MY02, and ginger extract (50 mg, 20% gingerols), marketed in France since January 2025 as Symbiosys® Stomalex.

A total of 198 adult patients with FD (Rome IV criteria, normal endoscopy) will be recruited in primary care and gastroenterology practices. After providing informed consent, eligible participants will receive one capsule per day for 8 weeks. The study involves two in-person visits (baseline and Week 8) and one telephone follow-up at Day 28.

The primary endpoint is the change in total PAGI-SYM score from baseline to Week 8.

Secondary endpoints include changes in PAGI-QoL scores, treatment adherence, use of concomitant therapies, evolution of lower gastrointestinal symptoms, global impressions of change from both patients (PGI-C) and physicians (CGI-I), and satisfaction ratings. An exploratory endpoint evaluates psychological impact using the Hospital Anxiety and Depression Scale (HADS). Safety endpoints include frequency and severity of adverse events.

This study will provide additional clinical evidence on the potential role of spore-forming probiotics combined with ginger extract as a complementary non-pharmacological approach to improve digestive symptoms and quality of life in patients with functional dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Adults (male or female) aged ≥18 years.
* Diagnosis of functional dyspepsia (FD) according to Rome IV criteria, with normal upper endoscopy including negative Helicobacter pylori test. Rome IV criteria define FD as the presence of one or more of the following symptoms: bothersome postprandial fullness, early satiety, epigastric pain, or epigastric burning, occurring at least 3 days per week during the last 3 months, with symptom onset at least 6 months prior to diagnosis.
* PAGI-SYM total score >1 at baseline.
* Ability to comply with study requirements and provide signed written informed consent before any study-related procedures.
* Ability to complete the patient diary and questionnaires, in the investigator's opinion (sufficient reading and language comprehension).
* For women of childbearing potential : Negative urine pregnancy test immediately before starting study product ; Agreement to use an approved method of contraception for the duration of the study, unless meeting criteria for menopause (≥12 months of spontaneous amenorrhea). Women of childbearing potential are defined as all women physiologically capable of becoming pregnant, including those whose career, lifestyle, or sexual orientation normally precludes heterosexual intercourse.
* Affiliation with a national health insurance or social security system.

Exclusion Criteria:

* Use within 2 weeks prior to baseline of treatments that could interfere with study evaluation, including Bacillus coagulans MY01, Bacillus subtilis MY02, ginger, peppermint, or antibiotics.
* Known allergy or hypersensitivity to any component of the investigational product.
* Contraindication or specific warning related to the investigational product, including use of anticoagulants.
* Use of immunosuppressive therapy within the last 3 months.
* Use of medications affecting gastrointestinal motility or sensitivity, including opioids, GLP-1 analogs, neuroleptics, antiemetics, or anticholinergics. (Stable antidepressant therapy allowed.)
* Significant changes in diet or physical activity within 2 weeks prior to baseline or anticipated during the study period.
* Active somatic or psychiatric disorder that could explain dyspeptic symptoms (e.g., active cancer, inflammatory disease). Stable use of one antidepressant is allowed for psychiatric indication.
* Active Helicobacter pylori infection.
* Predominant symptoms of gastroesophageal reflux disease (GERD) or irritable bowel syndrome (IBS).
* Functional diarrhea or functional constipation as defined by Rome IV criteria.
* History of abdominal surgery within the past year, except appendectomy, cholecystectomy, inguinal hernia repair, or splenectomy.
* Pregnant or breastfeeding women.
* Individuals under legal guardianship or curatorship.
* Participation in another interventional clinical trial and receipt of an investigational product within 30 days prior to baseline.
* Any acute or chronic medical or psychiatric condition that, in the investigator's judgment, could interfere with study assessments, including but not limited to severe hepatic or renal insufficiency, immunodeficiency, or substance abuse (alcohol or drugs).
* Any personal condition or circumstance that, in the investigator's judgment, would make full participation in the study unlikely or impossible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in PAGI-SYM total score from baseline to Week 8 | Baseline (Day 0) and Week 8 (Day 56 ± 3 days)
  The Patient Assessment of Gastrointestinal Symptom Severity Index (PAGI-SYM) is a validated questionnaire assessing severity of upper gastrointestinal symptoms. Total score ranges from 0 (none) to 5 (very severe). A decrease indicates symptom improvement.

SECONDARY OUTCOMES:
Change in Patient Assessment of Upper Gastrointestinal Symptom Severity Index (PAGI-SYM) Scores During Follow-up | Baseline, Weeks 2, 4, 6, and 8
  The PAGI-SYM (Patient Assessment of Upper Gastrointestinal Symptom Severity Index) is a validated patient-reported questionnaire assessing upper gastrointestinal symptoms. It includes 20 items scored on a 6-point Likert scale from 0 to 5 (0 = none, 5 = very severe). Subscale scores and the total score are calculated as the mean of completed items. Higher scores indicate worse symptom severity. A decrease from baseline reflects clinical improvement.
Change in Patient Assessment of Upper Gastrointestinal Quality of Life (PAGI-QoL) Total Score | Baseline, Week 4, and Week 8
  The PAGI-QoL (Patient Assessment of Upper Gastrointestinal Quality of Life) is a validated patient-reported questionnaire measuring quality of life in functional dyspepsia. It includes 30 items, each scored on a 6-point Likert scale from 0 to 5. Subscale and total scores are calculated as the mean of completed items. Total score range: 0 (lowest quality of life) to 5 (highest quality of life). Higher scores reflect better quality of life.
Patient adherence to study product assessed by patient diary | Week 4, and Week 8
  Adherence will be assessed using a patient diary in which participants record daily intake of the study product. Adherence will be expressed as the proportion of days with documented capsule intake relative to the total number of days.
Use of concomitant medications for dyspeptic symptoms | 2 months prior to inclusion and during study period (8 weeks)
  Proportion of patients using additional treatments for FD.
Evolution of lower gastrointestinal symptoms | Baseline and Week 8
  Change in presence/absence of symptoms compared to baseline.
Patient's Global Impression of Change (PGI-C) | Week 8
  The PGI-C (Patient's Global Impression of Change) is a self-reported 7-point Likert scale evaluating the patient's perception of change in health status since baseline. The scale ranges from 1 to 7, where 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. Lower scores (1-3) indicate clinical improvement, 4 indicates stability, and higher scores (5-7) indicate worsening.
Clinical Global Impression of Improvement (CGI-I) | Week 8
  The CGI-I (Clinical Global Impression of Improvement) is a physician-rated 7-point Likert scale assessing global improvement of the patient's condition compared with baseline. The scale ranges from 1 to 7, where 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse. Lower scores (1-3) indicate improvement, 4 indicates stability, and higher scores (5-7) indicate worsening.
Patient satisfaction with study product | Week 8
  5-point Likert scale (1 = not at all satisfied; 5 = very satisfied).
Physician satisfaction with study product | Week 8
  5-point Likert scale (1 = not at all satisfied; 5 = very satisfied).
Exploratory: Change in Hospital Anxiety and Depression Scale (HADS) score | Baseline and Week 8
  Evaluates impact on anxiety and depression. Total score ranges 0-21 per domain; higher scores indicate greater severity.
Safety and tolerability (Adverse Events) | From consent signature to Week 8 (end of study)
  Number, severity, and relationship of adverse events (AE) and serious adverse events (SAE).
Patient adherence to study product assessed by capsule count | Week 4 and Week 8
  Adherence will be assessed by counting the number of remaining capsules at study visits. Adherence will be expressed as the proportion of capsules taken relative to the number of capsules dispensed.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume GOURCEROL, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- Gerard DASSA, Istres, France